CLINICAL TRIAL: NCT02111356
Title: Quantative Analysis of Functional Changes by the Pinhole Glasses
Brief Title: Determine Functions of Pinhole Glasses on the Eyes
Acronym: PH001
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Principal Investigator, WonSoo Kim, WonSoo Kim, Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PH-001
Record Dates: First submitted 2014-04-04; First posted 2014-04-11 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Vision, Ocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pinhole glasses (Experimental): All subjects perform ophthalmic examinations before and after the pinhole glasses (Trayner Pinhole Glasses, Trayner Glasses, U.K.)
  Interventions: Device: Phinhole glasses

INTERVENTIONS:
Device: Phinhole glasses — Wearing the pinhole glasses (Trayner Pinhole Glasses, Trayner Glasses, U.K.)

SUMMARY:
Pinhole glasses which is using pinhole effect may induce a functional change on the eyes, including Distance and near visual acuity(DVA, NVA), Pupil size, DOF, Accomodative amplitude, CS, Visual field(VF), Stereopsis.

ELIGIBILITY:
Inclusion Criteria:

* Age : between 20 and 50 years old
* Visual acuity : correctable distant and near visual acuity by glasses up to 20/20
* Others : Normal intraocular pressure, optic discs with a healthy appearance, and normal ocular alignment.

Exclusion Criteria:

* History of systemic or topical medication that might affect accommodation
* Others : Corneal pathologic features, previous ocular surgery, glaucomatous optic discs, glaucoma, cataracts of grade II or greater, vitreous opacity, or retinal abnormalities that might limit the accuracy of test.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Distance and near visual acuity(DVA, NVA) | Change from baseline at 1 week
  Check distance(4m) and near(40cm) visual acuity using Snellen chart, Visual Acuity chart 2000, respectively.
  At 1 week, cheked with wearing the pinhole glasses (Trayner Pinhole Glasses, Trayner Glasses, U.K.)

SECONDARY OUTCOMES:
Pupil size | Change from baseline at 1 week
  Check the pupil size using WASCA Analyzer(Carl Zeiss Meditec, Germany)
Depth of focus | Change from baseline at 1 week
  Check with 4m Snellen chart.
  At 1 week, cheked with wearing the pinhole glasses (Trayner Pinhole Glasses, Trayner Glasses, U.K.)
Accomodation | Change from baseline at 1 week
  check by Donder's push-up method. The subject was instructed to view the target letter (20/20 reduced Snellen number), which initially was positioned at approximately 40 cm. The target then was moved progressively closer to the patient's eye at approximately 5 cm per second until the subject noticed the target starting to blur.
  At 1 week, cheked with wearing the pinhole glasses (Trayner Pinhole Glasses, Trayner Glasses, U.K.)
Visual field | Change from baseline at 1 week
  Humphrey Visual Field Analyzer (Carl Zeiss Meditec, Inc., Dublin, CA, USA) using a 30-2 Swedish Interactive Threshold Algorithm
  At 1 week, cheked with wearing the pinhole glasses (Trayner Pinhole Glasses, Trayner Glasses, U.K.)
Contrast sensitivity | Change from baseline at 1 week
  CSV-1000E Contrast Testing Instrument (VectorVision, Dayton, OH, USA) at 2.5m distance under the standard brightness (85 cd/m2)
  At 1 week, cheked with wearing the pinhole glasses (Trayner Pinhole Glasses, Trayner Glasses, U.K.)
Stereopsis | Change from baseline at 1 week
  Randot Stereotest (Stereo Optical Co, Chicago, Illinois, USA)
  At 1 week, cheked with wearing the pinhole glasses (Trayner Pinhole Glasses, Trayner Glasses, U.K.)

CONTACTS AND LOCATIONS:
Overall Officials: WonSoo Kim, M.D., Principal Investigator — Ophthalmology, Chung Ang University Hospital
Locations (1):
- Department of Ophthalmology, Chung-Ang University School of Medicine, Chung-Ang University Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim WS, Park IK, Chun YS. Quantitative analysis of functional changes caused by pinhole glasses. Invest Ophthalmol Vis Sci. 2014 Aug 12;55(10):6679-85. doi: 10.1167/iovs.14-14801. PMID 25118263